CLINICAL TRIAL: NCT02717819
Title: A Protein-enriched, Milk-based Supplement to Counteract Sarcopenia in Acutely Ill Geriatric Patients Offered Resistance Exercise Training During and After Hospitalisation - a Double-blinded, Randomized Controlled Trial
Brief Title: The Importance of Additional Protein to Benefit More From Training During and After Hospitalization
Acronym: PEPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forskningsenheden (Other)
Collaborators: University of Copenhagen (Other); The Danish Dairy Research Foundation, Denmark (Other); Arla Foods (Industry); Glostrup University Hospital, Copenhagen (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Forskningsenheden, Dietetics and Clinical Nutrition Research Unit, Copenhagen University Hospital at Herlev
Organization: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EFFECT.PEPOP.2016; H-16018240 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Muscular atrophy; Frailty; Acute illness; Ageing; Protein supplementation; Whey protein; Resistance training; Strength training
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Frailty | interventions — Proteins; Whey Proteins; Resistance Training; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training and protein (Experimental): Daily supervised resistance training offered while hospitalized, and encouragement of self-training 4 times per week for duration of 12 weeks after discharge (standardized training program, which will be monitered). Daily intake of 2 x 125 ml protein-enriched, milk-based supplements (whey protein), in the same period (additional ~25 g protein and 1953 kJ per day). Daily vitamin D supplements.
  Interventions: Dietary Supplement: Protein; Other: Resistance training; Dietary Supplement: Vitamin D
- Resistance training and placebo (Placebo Comparator): Daily supervised resistance training offered while hospitalized, and encouragement of self-training 4 times per week for duration of 12 weeks after discharge (standardized training program, which will be monitered). Daily intake of 2 x125 ml iso-energetic placebo-supplements, in the same period. Daily vitamin D supplements.
  Interventions: Dietary Supplement: Placebo; Other: Resistance training; Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Protein — Daily intake of supplement
  Other Names: Protein-enriched, milk-based supplement (whey protein)
  Arms: Resistance training and protein
Dietary Supplement: Placebo — Daily intake of supplement
  Other Names: Iso-energetic placebo-supplement (no protein)
  Arms: Resistance training and placebo
Other: Resistance training — Resistance training (offered daily while hospitalized, and encouragement of 4 x/week as self-training after discharge)
Dietary Supplement: Vitamin D — Aiming at a dose of 20 ug/day. 20 ug/day will be handed out to study participants who do not get vitamin D supplements from the hospital while admitted and to those who are not already taking vitamin D supplements themselfes e.g. as part of a combination tablet.

SUMMARY:
The purpose of the study is to investigate if an increased protein intake, in the form of a protein-enriched, milk-based supplement, can enhance the beneficial effect of resistance training, offered during hospitalization and 12 weeks post discharge, in older patients. This will in part be evaluated from measures of muscle strength, muscle mass and physical functioning. Also, the study population's acceptance of the intervention product will be assessed along with measures related to 'cost-effectiveness'.

A sub-study will be performed in a sub-group (n=30) to investigate if bio-impedance analysis (BIA) correlates with Dual-Energy X-ray absorptiometry (DXA) at single time points, and to see if it is possible to track changes in lean body mass. In addition, the reliability of the bio-impedance analyzer will be evaluated.

Also, the prevalence and classification of sarcopenia will be assessed at baseline, and correlations to nutritional status will be investigated (n=120).

DETAILED DESCRIPTION:
Main study:

The study design is a block randomised, double-blind, placebo-controlled, multicentre intervention study. A total of 120 hospitalized older adults, above 70 years, will be recruited consecutively from the medical departments of three Hospitals in the Capital Region of Denmark (n=40 each place).

Participants will be randomized into two groups - one group receives protein-enriched, milk-based supplements and the other group receives iso-energetic placebo products. Both groups participate in the same standardized resistance training program, and will be blinded to the supplement content. One training session consists of three exercises of the lower extremities (3 sets of 10 repetitions, pursuing an intensity of 8-12 repetition maximum (RM)). While admitted, supervised resistance training is offered daily. After discharge, the participants are encouraged to perform the same program as self-training four times per week.To ensure progression (or regression if necessary) the participants receive follow-up home visits by a physiotherapist, and thus after discharge the participants are closely monitored. All participants, irrespective of allocation, will get a daily vitamin D supplement.

The study duration for each participant starts while admitted to hospital and lasts until 12 weeks after discharge. Endpoint assessments will be performed at baseline (> 72-h after admission to hospital), after discharge (> 72-h) and 12 weeks (± 2 days) after discharge. A few endpoints will be collected during follow-up (6 months post intervention). Data will be collected by study investigators blinded to the allocation of the participants.

Sub-study: 'Validation of a portable bio-impedance analyzer in a population of older adults ≥ 70 years for the assessment of muscle mass and changes in muscle mass over time' A sub-study will be performed to investigate if the portable InBody-230 BIA correlate with DXA at single time points in 30 hospitalized older people ≥ 70 years, and to see if it is possible to track changes in LBM during the 12-week intervention. Total LBM, total fat mass, and percent LBM will be measured and compared as well as appendicular and trunk LBM. In addition, the reliability of the portable bio-impedance analyzer will be evaluated by assessing the degree of agreement between two subsequent measurements. In continuation of recruitment to the primary study, a subset of participants (n=30) will be asked if they want to participate in this sub-study, irrespective of their allocation in the main study. The measurements are going to be performed twice, while hospitalized and 12 weeks after discharge (± 5 days).

Sub-study: 'Prevalence of sarcopenia and investigation of the relationship between nutritional status and the EWGSOP conceptual stages for sarcopenia in hospitalized older patients > 70 years'.

The prevalence and classification of sarcopenia among Danish hospitalized older patients ≥ 70 years old (n=120) will be evaluated, according to the EWGSOP definition (Hand-grip-strength, 4-m gait speed, Bio-Impedance analysis). Also, examination of the relationship between measurements of nutritional status and the EWGSOP stages for sarcopenia (i.e. no sarcopenia, pre-sarcopenia, sarcopenia and severe sarcopenia) will be assessed at baseline. Nutritional status will be assessed according to BMI (< 18.5, 18.5-20.5, 20.5-25, > 25), Mini Nutritional Assessment (MNA) (no MN, risk of MN, MN), Malnutrition Universal Screening Tool (MUST) (low risk of MN, medium risk of MN, high risk of MN), and NRS-2002 (no MN, mild MN, moderate MN, severe MN)

Results will be communicated to the general population and published in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 70 years old
* Able to speak and understand Danish
* Expected length of stay > 3 days (evaluated by medical staff at department)
* Ability to stand independently without walking aids
* Admitted to the medical departments of Gentofte or Herlev Hospital or Rigshospitalet-Glostrup

Exclusion Criteria:

* Active cancer
* Renal insufficiency (eGFR < 30 mL/min/1.73m2)
* Cognitive impairment (not able to comprehend the purpose of the study/give informed consent)
* Terminal disease
* Exclusively receiving enteral or parenteral nutrition
* Milk/lactose allergy or intolerance
* Planning to lose weight/go on a special diet
* Planned transfer to other hospitals/departments
* Pacemaker/other implanted electrical stimulants (due to Bio-Impedance Analysis (BIA) measurements)
* Not being able to lie still in seven minutes (only an exclusion criteria in the sub-study)
* Withdrawal criteria: Death during admission (does not apply to subsequent admissions)
* Withdrawal criteria: Discharge/transfer from the medical department before the intervention has started

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Change in 30-s chair stand performance | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Number of stand-ups from a chair in 30 seconds (modified version, help from armrests are allowed).

SECONDARY OUTCOMES:
Total lean body mass | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Lean body mass (kg and percent) evaluated by bio-impedance analysis (portable, dual-frequency, 8-Point Tactile Electrode System).
Appendicular lean body mass | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Appendicular lean body mass (kg and percent) evaluated by bio-impedance analysis (portable, dual-frequency, 8-Point Tactile Electrode System).
Trunk lean body mass | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Trunk lean body mass (kg and percent) evaluated by bio-impedance analysis (portable, dual-frequency, 8-Point Tactile Electrode System).
Change in hand grip strength | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Isometric hand grip strength (kg) (Saehan Medical digital dynamometer, 2012).
Change in 4 m gait speed | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  The time used for walking 4 m (m/s and s )
Change in Activities of daily living (ADL) | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Use of Barthel-100
Change in mobility | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Use of De Morton Mobility Index (DEMMI)
Change in cognitive functioning | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Use of Mini Mental State Examination (MMSE)
Use of home care | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Interview: (yes/no)
Residence | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Interview: (own home, nursing home/assisted living facility, 24-hour rehabilitation facility)
Use of gait aid | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Interview: yes/no/cannot walk and registration of specific gait help
Length of hospital stay (LOS) | Day of discharge (from hospital)
  The in-hospital intervention period (date of recruitment until date of discharge) (days)
Readmission to hospital | From discharge until 12 weeks post discharge, and 6 months post discharge
  Frequency (number)
Length of total hospital stay for readmissions | From discharge until 12 weeks post discharge, and 6 months post discharge
  Total length (days).
Mortality | From discharge until 12 weeks post discharge, and 6 months post discharge
  Mortality (yes/no)
Change in health related Quality of life | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Questionnaire: Euroqol EQ-5D-3L
Change in Body weight | Baseline (admission to hospital), within 3 days of discharge, and 12 weeks after discharge
  Measured to the nearest 0.1 kg using a calibrated scale
Study population acceptance of product | 12 weeks post discharge
  Self-administered evaluation-questionnaire

OTHER OUTCOMES:
Lean body mass (sub group n=30) | Baseline (while admitted to hospital) and 12 weeks post discharge
  Lean body mass (total, appendicular, and trunk) evaluated by whole-body dual energy x-ray absorptiometry (DXA)-scanning.
Fat mass (sub group n=30) | Baseline (while admitted to hospital) and 12 weeks post discharge
  Total mass. Evaluated by whole-body dual energy x-ray absorptiometry (DXA)-scanning and bio-impedance analysis (BIA).
Reliability of bio-impedance analyzer in sub-group (n=30) | Baseline (while admitted to hospital)
  Degree of agreement between two subsequent measurements.
Prevalence of sarcopenia | Baseline (while admitted to hospital)
  According to the EWGSOP definition (yes/no).
Classification of sarcopenia | Baseline (while admitted to hospital)
  According to the EWGSOP definition (pre-sarcopenia, sarcopenia, and severe sarcopenia).
Nutritional status - Body mass index (BMI) | Baseline (while admitted to hospital)
  According to BMI (kg/m2) (< 18.5, 18.5-20.5, 20.5-25, > 25)
Nutritional status - Mini Nutritional Assessment (MNA) | Baseline (while admitted to hospital)
  According to Mini Nutritional Assessment (MNA) (no malnutrition, risk of malnutrition, malnutrition).
Nutritional status - Malnutrition Universal Screening Tool (MUST) | Baseline (while admitted to hospital)
  According to Malnutrition Universal Screening Tool (MUST) (low risk of MN, medium risk of MN, high risk of MN)
Nutritional status - Nutritional Risk Screening 2002 (NRS-2002) | Baseline (while admitted to hospital)
  According to Nutritional Risk Screening 2002 (NRS-2002) (no MN, mild MN, moderate MN, severe MN).
Energy intake | 4 days while admitted to hospital, or shorter if discharged
  Daily registration schemes with pre-printed hospital foods and drinks (energy, kJ/kg).
Protein intake | 4 days while admitted to hospital, or shorter if discharged
  Daily registration schemes with pre-printed hospital foods and drinks (protein, g/kg).
Energy intake | From discharge until 12 weeks post discharge
  Dietary interviews x 4 (24-h recall interviews) (energy, kJ/kg).
Protein intake | From discharge until 12 weeks post discharge
  Dietary interviews x 4 (24-h recall interviews) (protein, g/kg).
Level of daily activity | From discharge until 12 weeks post discharge
  Activity interviews x 4 (recall interviews for the previous week)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, DMSc, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital Gentofte, Gentofte Municipality
  - Rigshospitalet-Glostrup, Glostrup Municipality
  - Copenhagen University Hospital Herlev, Herlev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gade J, Beck AM, Andersen HE, Christensen B, Ronholt F, Klausen TW, Vinther A, Astrup A. Protein supplementation combined with low-intensity resistance training in geriatric medical patients during and after hospitalisation: a randomised, double-blind, multicentre trial. Br J Nutr. 2019 Nov 14;122(9):1006-1020. doi: 10.1017/S0007114519001831. PMID 31337448
- [Derived] Gade J, Beck AM, Bitz C, Christensen B, Klausen TW, Vinther A, Astrup A. Protein-enriched, milk-based supplement to counteract sarcopenia in acutely ill geriatric patients offered resistance exercise training during and after hospitalisation: study protocol for a randomised, double-blind, multicentre trial. BMJ Open. 2018 Feb 1;8(2):e019210. doi: 10.1136/bmjopen-2017-019210. PMID 29391380